CLINICAL TRIAL: NCT00215995
Title: A Phase II Study of Cisplatin and Irinotecan Induction Chemotherapy, Followed by ZD 1839 (IRESSA) in Adult Patients With Surgically Unresectable and/or Metastatic Esophageal or Gastric Carcinomas
Brief Title: Cisplatin and Irinotecan Chemotherapy, Followed by ZD 1839 (Iressa) in Patients With Esophageal or Gastric Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13426; USFIRB#101525
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2007-05

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: esophageal cancer; esophagogastric cancer; gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Cisplatin; Irinotecan; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin, Irinotecan and ZD1839 (Experimental): As outlined in Detailed Description.
  Interventions: Drug: Cisplatin; Drug: Irinotecan; Drug: ZD 1839

INTERVENTIONS:
Drug: Cisplatin — As outlined in Detailed Description
  Other Names: Platinol; Platinol-AQ
Drug: Irinotecan — As outlined in Detailed Description
  Other Names: Camptosar
Drug: ZD 1839 — As outlined in Detailed Description
  Other Names: Iressa

SUMMARY:
This study is for patients with esophageal, esophagogastric, or gastric cancer that has spread to other parts of the body. The purpose of this study is to test the safety and effectiveness of a new experimental drug called ZD 1839 following initial therapy with two other chemotherapy drugs, called Irinotecan (CPT-11) and Cisplatin.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multicenter Phase II study designed to evaluate tumor response rates in patients with surgically unresectable and/or metastatic esophageal, esophagogastric, and gastric adenocarcinoma or squamous carcinoma. Study schema is as follows. Patients will receive Irinotecan and Cisplatin on days 1 and 8 every 21 days for a maximum of 6 cycles of therapy. This is then followed by ZD 1839 (Iressa), which is an oral pill taken once daily. During the Iressa phase, patients will be evaluated every 6 weeks. This includes labs, CT scans and physical examination. The exploratory objective of the study is to examine the correlation between epidermal growth factor receptor (EGFR) expression and radiographic response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of esophageal carcinoma (squamous or adenocarcinoma) or gastric adenocarcinoma.
* Surgically unresectable disease and/or metastatic disease.
* No prior chemotherapy therapy.
* Life expectancy > 12 weeks.
* Patients must have the ability to take and retain oral medications.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Karnofsky Performance Status [KPS] ≥50%).
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria and computerized tomographic scan performed within 28 days prior to registration.
* Organ system function assessed within 7 days prior to registration and within the following parameters:

  * Absolute neutrophil count ≥1500/mL;
  * Platelet count ≥100,000/mL;
  * Hemoglobin level ≥10.0 gm/dL;
  * Serum creatinine ≤1.5 x IULN (Institutional Upper Limits of Normal); OR Measured creatinine clearance ≥60 mL/min;
  * AST (SGOT) or ALT (SGPT) ≤ 2.5 x IULN (unless the liver is involved by tumor, in which case it must be ≤5.0 x IULN);
  * Total bilirubin ≤1.5 x IULN.
* Understanding of the subject of the potential and unknown teratogenic risk, as well as their willingness to practice birth control. Should a pregnancy occur while a subject, either father or mother, is receiving study medication, the subject should inform the doctor immediately.
* Aged 18 years or older
* Provision of written informed consent
* For patients with locally advanced disease, subjects must be evaluated by a radiation oncologist prior to study entry, and judged that radiation therapy is not indicated in the subjects therapy.

Exclusion Criteria:

* Prior treatment with EGFR-inhibiting agents, chemotherapy, or radiotherapy for esophagogastric carcinomas.
* Patients must not be receiving any other investigational agents. Use of erythropoietin is allowable. Secondary prophylaxis with granulocyte colony stimulating factor (G-CSF) (Filgrastim) is allowable. The use of granulocyte-macrophage colony stimulating factor (GM-CSF) (Sargramostim) is not allowed on this protocol.
* Uncontrolled brain metastases.
* Patients must not have uncontrolled intercurrent illness at the time of registration including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina, pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not have current New York Heart Association Class III or IV heart disease.
* Known human immunodeficiency virus (HIV) infection.
* Pregnant or breast-feeding women.
* Patients who have had prior malignancies, except non-melanoma skin cancer (basal or squamous cell carcinoma) are not eligible for this study; unless greater than 5 years has passed since the event.
* Known severe hypersensitivity to ZD 1839 or any of the excipients of this product.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St. John's Wort.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.
* Incomplete healing from previous oncologic or other major surgery.
* Serum creatinine level greater than Common Toxicity Criteria (CTC) grade 2.
* Any evidence of clinically active interstitial lung disease. Subjects with chronic stable radiographic changes who are asymptomatic need not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Desired Response | 48 Months
  Response rate

SECONDARY OUTCOMES:
Duration of Participants' Desired Response | 48 Months
  Response duration in months
Participants' Time to Disease Progression | 48 Months
  Time to progression in months
Number of Participants With Overall Survival | 48 Months
  Overall survival from first participant On Treatment to last participant Off Study

CONTACTS AND LOCATIONS:
Overall Officials: Chris Garrett, MD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (3):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - University of Puetro Rico Cancer Center, San Juan

REFERENCES:
- See also: Moffiitt Cancer Center Clinical Trials website — http://www.moffitt.org